CLINICAL TRIAL: NCT02149472
Title: Towards Better Prognostic and Diagnostic Strategies for Haemostatic Changes During Major Obstetric Haemorrhage
Acronym: TeMpOH-2
Status: Completed | Type: Observational
Sponsor: Sanquin-LUMC J.J van Rood Center for Clinical Transfusion Research (Other)
Collaborators: Leiden University Medical Center (Other); Erasmus Medical Center (Other); Isala (Other)
Responsible Party: Sponsor
Other Study IDs: NL.46563.058.13; P13.246 (Other: Leiden University Medical Center (LUMC))
Record Dates: First submitted 2014-05-12; First posted 2014-05-29 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be drawn for conventional haemostatic parameters and ROTEM profiles. Remaining plasma will be frozen and stored for further evaulation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women with PPH: All pregnant women in participating hospitals are asked for their informed consent (n = 9.500). All women will complete a bleeding score generating questionnaire during their pregnancy. Only from women developing postpartum haemorrhage > 1000 cc blood samples will be drawn (n = 600).

SUMMARY:
Major obstetric haemorrhage (MOH) remains a cause of significant maternal morbidity and mortality worldwide. By identifying women with a higher a priori risk of major haemorrhage during their pregnancy or early during postpartum haemorrhage extra measures to prevent MOH can be taken.

In this study the investigators aim to identify haemostatic parameters that during the course of haemorrhage are responsible for the on-going towards major bleeding. By doing this, cut-off points can be defined for future interventions aiming to stop this bleeding process in an early stage. Traditional coagulation parameters are currently not useful for clinical decision making, because of long turn around times. Therefore the added value of available coagulation 'point of care' tests will be evaluated during obstetric haemorrhage.These Point-of-Care (POC) tests could lead to a goal-directed haemostatic therapy for obstetric haemorrhage.

A cohort of 9.500 pregnant women will be followed during their pregnancy and delivery. From all women a bleeding score will be obtained during their pregnancy by means of a validated questionnaire. The predictive value of this bleeding score for the occurrence of major obstetric haemorrhage will be evaluated.

If postpartum haemorrhage develops (blood loss) > 1000 cc, blood samples will be drawn for conventional haemostatic parameters and ROTEM profiles. The pathway between minor bleeding and major bleeding will be elucidated. Interchangeability and comparability of conventional haemostatic parameters and ROTEM profiles will also be evaluated.

The overall goal of the investigators is becoming more able to predict major obstetric haemorrhage in an early stage of postpartum haemorrhage and define thresholds for goal-directed hemostatic therapies.

DETAILED DESCRIPTION:
See 'brief summary'

ELIGIBILITY:
Inclusion Criteria:

- Pregnancy, gestation age > 24 weeks

Exclusion Criteria:

* Age < 18
* Adults incapable of giving informed consent
* Gestational age < 24 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All pregnant women in participating hospitals are asked for their informed consent (n = 9.500). All women will complete a bleeding score generating questionnaire duing their pregnancy. Only from women developing postpartum haemorrhage > 1000 cc blood samples will be drawn (n = 600) during the course of postpartum haemorrhage for evaluation of changes in haemostatic parameters and ROTEM profiles.
  3 months postpartum a nested case cohort study will be performed to compare the incidences of underlying bleeding disorders in the haemorrhage and non-haemorrhage group. This outcome will also be related to the obtained bleeding scores during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 1649 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Early haemostatic predictors of major obstetric haemorrhage | Postpartum haemorrhage within the 24 hrs hours after childbirth
  During early postpartum haemorrhage changes in hemostatic parameters leading to major obstetric haemorrhage will be identified. Conventional hemostatic parameters and ROTEM profiles will be studied.

SECONDARY OUTCOMES:
Evaluation of ROTEM-based MOH prediction scores as alternative to traditional haemostatic parameters | Postpartum haemorrhage within first 24 hrs after childbirth
Incidence of underlying bleeding disorders in patients with MOH | 3 months postpartum
Predictive value bleeding score in pregnancy for MOH | Third trimester of pregnancy - 24 hours postpartum

CONTACTS AND LOCATIONS:
Overall Officials: J G van der Bom, Prof, MD,PhD, Principal Investigator — LUMC and Center for Clinical Transufion Research Sanquin
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tahitu M, Ramler PI, Gillissen A, Caram-Deelder C, Henriquez DDCA, de Maat MPM, Duvekot JJ, Eikenboom J, Bloemenkamp KWM, van den Akker T, van der Bom JG. Clinical value of early assessment of hyperfibrinolysis by rotational thromboelastometry during postpartum hemorrhage for the prediction of severity of bleeding: A multicenter prospective cohort study in the Netherlands. Acta Obstet Gynecol Scand. 2022 Jan;101(1):145-152. doi: 10.1111/aogs.14279. Epub 2021 Nov 3. PMID 34729767